Document: TDOC-0055987

Status: Effective

Version: 1.0; CURRENT; Most-Recent; Effective

Effective Date: 24-Apr-2019

**Short Title** 

# ClarVista CP-00004

Long Title

# A PROSPECTIVE, MULTI-CENTER STUDY TO EVALUATE THE SAFETY AND PERFORMANCE OF THE EXCHANGEABLE CLARVISTA HARMONI™ MODULAR TORIC INTRAOCULAR LENS SYSTEM FOR THE TREATMENT OF PRE-EXISTING CORNEAL ASTIGMATISM AND APHAKIA FOLLOWING CATARACT

# 1 TITLE PAGE

Protocol Number: ClarVista CP-00004 / NCT03050697

Medical Specialty: Surgical

Project Name /Number: NA

Sponsor Name & Address: CLARVISTA MEDICAL, INCORPORATED

26800 ALISO VIEJO PARKWAY, SUITE 120

ALISO VIEJO, CA 92656 PHONE +001 949 916-5412 FAX +001 949 916-5412

Test Article(s) / Product(s): ClarVista HARMONI® Modular Toric Intraocular Lens

System

**Document:** TDOC-0055987

Status: Effective


CLARVISTA MEDICAL

Effective Date: 24-Apr-2019





A Prospective, Multi Center Study to Evaluate the Safety and Performance of the Exchangeable ClarVista Harmoni™ Modular Toric Intraocular Lens System For The Treatment Of Pre Existing Corneal Astigmatism and Aphakia Following Cataract Surgery

Protocol Number #CP-00004 REV.01

Sponsor ClarVista Medical, Incorporated

26800 ALISO VIEJO PARKWAY, SUITE 120

ALISO VIEJO, CA 92656 PHONE +001 949 916-5412 FAX +001 949 916-5412

Original Version Date (Rev.01) 06 June 2016

This cinical investigation is being conducted in accordance with 21 CFR Parts 11, 50, 54, 56, and 812, SO 14155 (2011) Cinical investigation of Medical Devices for Human Subjects, SO 11979 7:2014 Ophthamic implants—intraocular enses—Part 7, : Cinical investigations (where applicable), ANS Z80 7 2013 Ophthamic Optics—intraocular Lenses (where applicable), CH GCPs, and applicable ocal regulations

#### CONFIDENTIAL

The information in this document is confident a and will not be disclosed to others without written authorization from ClarV stall Medical, except to the extent necessary to obtain informed consent from persons involved in the clinical study or their legal guardians, or for discussions with local regulatory authorities, institutional review boards (RB), Ethics Committees (EC) or persons participating in the conduct of the trial

Document: TDOC-0055987

Status: Effective


#### PROTOCOL # CP-00004 REV.01

#### CLARVISTA MEDICAL

Effective Date: 24-Apr-2019

# **PROTOCOL CONTACTS**

## Sponsor

ClarVista Medical 26800 Aliso Viejo Parkway, Suite 120 Aliso Viejo, CA 92656

Ph: +001.949.916.5412







Rev 01, 06 June 2016 

Print Date: Printed By:

Document: TDOC-0055987

Status: Effective


CLARVISTA MEDICAL

Effective Date: 24-Apr-2019

PROTOCOL # CP-00004 REV.01

# PROTOCOL APPROVAL

A Prospect ve, Mu t -Center Study to Eva uate the Safety and Performance of the C arV sta HARMONI® Modu ar Tor c Intraocu ar Lens System for the Treatment of Pre-Ex st ng Cornea Ast gmat sm and Aphak a Fo ow ng Cataract Surgery

The fo ow ng nd v dua s approve Protoco #CP-00004 Rev.01 dated 6 June 2016. Any changes to th s vers on of the protoco must have an amendment or adm n strat ve etter.

C arV sta Approva s:



**Document:** TDOC-0055987

Status: Effective


CLARVISTA MEDICAL

Effective Date: 24-Apr-2019

PROTOCOL # CP-00004 REV.01

#### STUDY ACKNOWLEDGEMENT

I understand this protoco contains information that is confident a and proprietary to ClarV sta Medical (ClarV sta).

I have read this protoco and agree that it contains a in the details necessary to conduct the study as described. I will follow this protoco in the conduct of the study and will make a reasonable effort to complete the study in the time noted.

I w prov de the contents of th s protoco to study staff under my d rect superv s on n order to conduct the study. I w d scuss th s nformat on w th the study staff to ensure they are fu y nformed about the study and the test art c e. I w prov de the contents of the protoco to the respons b e Eth cs Comm ttee. These d sc osures may be made; prov d ng the contents are not used n any other c n ca study and they are not d sc osed to any other person or ent ty w thout pr or wr tten consent from C arV sta. Th s cond t on does not app y to d sc osure required by government regulations or laws; however, I agree to give prompt not ce to C arV sta of any such d sc osure.

I understand the study may be term nated or enroment suspended at any time by C arV sta, with or without cause, or by me if it becomes necessary to protect the interests of the study subjects.

Any add t ona  $\,$  nformat on added to th s protoco  $\,$  s a so conf dent a  $\,$  and propr etary to C arV sta and must be treated  $\,$  n the same manner as the contents of th s protoco  $\,$ .

| Pr nted Name of Pr nc pa Invest gator | |
|---------------------------------------|----------|
| Invest gator S gnature | <br>Date |

Protoco # CP-00004 Rev.01

Date: 06 June 2016

# Document: TDOC-0055987 Ve


Status: Effective

#### PROTOCOL # CP-00004 REV.01

#### CLARVISTA MEDICAL

Effective Date: 24-Apr-2019

| Table | e of ( | Conte | nts | |
|---|---|---|---|---|
| | 1 | | | |
| | | | A CENTER | |
| | | | MENT | |
| | | | is | |
| 1.0 INT | RODUCT | ION | | 15 |
| 3.0 STU | DY DES: | | TOUGHT STUDY | |
| | 3 2 | | T ON O THE STUDY<br>PO ULAT ON | 17 |
| | 3 2 | | | |
| | | 3 2 1 | nc us on Cr ter a | 17 |
| | | 3 2 2 | Exc us on Cr ter a Pr or to Surgery | 18 |
| | | 3 2 3 | D scont nuat on Cr ter a Dur ng Surgery | 19 |
| | 3 3 | STUDY \ | √s ts | 20 |
| | | 3 3 1 | Pre Operat ve V s t – Screen ng/Base ne (Day 90 to Day 0) | 20 |
| | | 3 3 2 | Day 0 V s t (Cataract Surgery and OL mp antat on) | 20 |
| | | 3 3 3 | Post Operat ve V s ts (Days 1 – 60) | 21 |
| | | 3 3 4 | 3 Month V s t (Day 80 100) | 21 |
| | | 3 3 5 | Unschedu ed V s ts | 2: |
| | | 3 3 6 | M ssed V s ts | 22 |
| 4.0 | STUDY | МЕТНО | DS | 22 |
| | 41 | | IED CONSENT | 22 |
| | 4 2 | Ass gni | MENT O SUBJECT DENT CAT ON | 22 |
| | 4 3 | SCREEN | FA LURE | 23 |
| | 4 4 | SUBJECT | T COM LET ON | 23 |
| | 4 5 | | T D SCONT NUAT ON | 23 |
| | 4 6 | | Follow U | 23 |
| | 4 7 | STUDY C | COM LET ON | 24 |
| | | 471 | Ear y Study Term nat on | 24 |
| | 4 8 | Concor | M TANT THERA ES | 24 |
| | | 481 | Concom tant Med cat on | 24 |
| | | 482 | Concom tant Procedures | 24 |
| - 0 | 4 9 | | COL DEV AT ONS | 25 |
| 5.0 | | | IALS | |
| | 5 1 | | TON O TEST ART CLE | 25 |
| | | 511 | nstruct ons for Use | 26 |
| | 5 2 | PACKAG | S NG AND LABEL NG | 26 |
| | 5 3 | Accoun | NTAB L TY | 26 |

Rev 01, 06 June 2016

Page **5** of **40** 


PROTOCOL # CP-00004 REV.01

# Document: TDOC-0055987


Effective Date: 24-Apr-2019

CLARVISTA MEDICAL

Status: Effective

| 5.0 | 5 4<br>Adve | | Mater als | 27<br>27 |
|---|---|---|---|---|
| | 61 | DE NT | | 27 |
| | | 611 | Adverse Event (AE) | 27 |
| | | 612 | Adverse Dev ce Effect (ADE) | 28 |
| | | 613 | Unant c pated Adverse Dev ce Effect (UADE) | 28 |
| | | 614 | Dev ce Def c enc es (DD) | 29 |
| | 6 2 | AE EVAI | LUAT ON | 29 |
| | | 621 | Eva uat on | 29 |
| | 6 3 | RE ORT | NG | 31 |
| | | 6 3 1 | On S te Exped ted Report ng | 31 |
| | | 6 3 2 | Off S te SAE Report ng | 32 |
| | | 6 3 3 | Report ng of Comp a nts for Anc ary Marketed Products | 32 |
| | | 6 3 4 | Adverse Events and Ser ous Adverse Events at Sub ect Ex t | 32 |
| | 6 4 | | Mon tor ng and Rev ew | 32 |
| .0 | | STUDY OUTCOMES | | |
| | 7 2 | | | |
| .0 | STATI<br>8 1 | | AETHODS | 33 |
| | 82 | | ES PO ULAT ONS | 34 |
| | | 821 | Safety Popu at on | 34 |
| | | 822 | mp anted Eye Popu at on | 34 |
| | | 823 | Per Protoco Popu at on | 34 |
| | 8 3 | STAT ST | CAL METHODS | 35 |
| | | 831 | Safety Outcomes | 35 |
| | | 832 | Performance Outcomes | 35 |
| .0 | | | MENT | |
| | 9 1 | | QUAL TY ASSURANCE | 37 |
| | | 911 | Data Mon tor ng | 37 |
| | 9 2 | | RETENT ON | 38 |
| 0.0 | K F F F i | RENCES | | |


Page **6** of **40** 

Printed By: Print Date:

Rev 01, 06 June 2016

**Document:** TDOC-0055987 **Version:** 1.0; CURRENT; Most-Recent; Effective

Status: Effective

#### PROTOCOL # CP-00004 REV.01

#### CLARVISTA MEDICAL

Effective Date: 24-Apr-2019

# **TABLE OF FIGURES**

| F GURE 1 | COHORT SCHEDULE | 10 |
|----------|-----------------------------------------------------|----|
| F GURE 2 | COHORT SCHEDULE | 17 |
| F GURE 3 | THE HARMON ™ MODULAR NTRAOCULAR LENS (HM OL) SYSTEM | 26 |

# LIST OF ABBREVIATIONS

| Abbreviation/Acronym | Term |
|----------------------|----------------------------------------------------|
| AE | Adverse Event |
| | Anter or Chamber Depth |
| | Adverse Dev ce Effect |
| AL | Ax a Length |
| | Amer can Nat ona Standards Inst tute |
| BCDVA | Best-Corrected D stance V sua Acu ty |
| CFR | Code of Federa Regu at ons |
| D | D opter |
| DD | Dev ce Def c enc es |
| DFE | D ated Fundus Exam nat on |
| EC | Eth cs Comm ttee |
| eCRF | E ectron c Case Report Form |
| ETDRS | Ear y Treatment D abet c Ret nopathy Study (Chart) |
| EtO | Ethy ene ox de |
| FDA | Un ted States Food and Drug Adm n strat on |
| GCPs | Good C n ca Pract ces |
| HIPAA | Hea th Insurance Portab ty and Accountab ty Act |
| HMTIOL | HARMONI™ Modu ar Tor c Intraocu ar Lens System |
| | Invest gator Brochure |
| | Informed Consent Form |
| ICH | Internat ona Conference on Harmon zat on |
| · | Ident f cat on |
| IDE | Invest gat ona Dev ce Exempt on |
| OA | ntraoperat ve Aberrometry |
| IOL | Intraocu ar Lens |
| | Intraocu ar Pressure |
| | Inst tut ona Rev ew Board |
| ISO | Internat ona Organ zat on for Standard zat on |
| | Keratometry |
| | Laser In-S tu Keratom eus s |
| | Man fest Refract on |
| | Man fest Refract on Cy nder |
| | Man fest Refract on Spher ca Equ va ent |
| | Neodym um:Yttr um-a um num-garnet |
| | Not Done |
| | R ght Eye |
| OS | Left Eye |


Status: Effective

#### PROTOCOL # CP-00004 REV.01

#### CLARVISTA MEDICAL

Effective Date: 24-Apr-2019

| OVD | Ophtha m c V scoe ast c Dev ce |
|-------|-----------------------------------|
| PCO | Poster or Capsu e Opac f cat on |
| PE | Pred ct on Error |
| PH | P nho e |
| PMA | Premarket Approva |
| PP | Per Protoco |
| PRK | Photorefract ve Keratectomy |
| RRE | Res dua Refract ve Error |
| SAE | Ser ous Adverse Event |
| SIA | Surg ca y Induced Ast gmat sm |
| SLE | S t Lamp Exam nat on |
| SOC | Standard of Care |
| SPK | Superf c a Punctate Kerat t s |
| SSI | Secondary Surg ca Intervent on |
| TRRE | Target Res dua Refract ve Error |
| UCDVA | Uncorrected D stance V sua Acu ty |
| US | Un ted States |
| VA | V sua Acu ty |

NOTE: The first occurrence of some abbreviations are not spelled out in the document (e.g. units of measure)


Status: Effective

CLARV STA MED CAL PROTOCOL CP 00004 Rev 01

Effective Date: 24-Apr-2019

# **PROTOCOL SYNOPSIS**

| Protocol Number | |
|---|---|
| | #CP-00004 Rev.01 |
| Title A Prospect ve, Mu t -Center Study to Eva uate the Safety and Perform the C arV sta HARMONI® Modu ar Tor c Intraocu ar Lens System Treatment Of Pre-Ex st ng Cornea Ast gmat sm and Aphak a Fo Cataract Surgery | |
| Regulatory Status | Phase 4 n CE countr es |
| | US - Pre-IDE |
| Investigational Device | C arV sta HARMON Modu ar Tor c ntraocu ar Lens System (HMT OL) |
| Objectives | A study to eva uate the safety and performance of the HMTIOL n pat ents w th pre-ex st ng cornea ast gmat sm. Spec f ca y, |
| | <ul> <li>To ref ne the A-constant (ens constant) of the HMTIOL.</li> <li>To eva uate the refract ve outcomes nc ud ng ast gmat sm correct on w th HMTIOL n pr mary cataract surgery.</li> <li>To eva uate ax a and rotat ona stab ty of the HMTIOL</li> </ul> |
| Number of Clinical Sites<br>and Study Subjects | Up to 200 enro ed and mp anted eyes from up to 10 nvest gat ona s tes. Approx mate y 20 eyes, a max mum of 30, w be enro ed from each nvest gator/surgeon. Enro ment w be mon tored as out ned n Samp e S ze sect on and adjusted accord ng y. |
| Study Duration | A subjects w part c pate n the study for up to 6 months (3 months pre-op w ndow p us 3 months fo ow up per od). Tota study durat on w be approx mate y 9 months. |
| Study Design | Prospect ve, mut-center c n ca study. A subjects w be seen for a Preoperat ve V st to capture base ne measurements. One or both eyes of each subject w undergo cataract surgery and be mp anted w th the HMTIOL. Eyes w th cornea ast gmat sm wh ch s w th n the d optr c range of the tor c IOL (1.50, 2.25 and 3.00D at the IOL p ane after adjust ng for Surg ca y Induced Ast gmat sm) may be mp anted w th the study dev ce. Fo ow up: |

**Document:** TDOC-0055987 **Version:** 1.0; CURRENT; Most-Recent, Effective

Status: Effective


Effective Date: 24-Apr-2019

| | 45 414 1 444 1 1044 1 6 |
|---|---|
| | 1 Day, 1 Week, 1 Month, and 3 Months fo ow ng cataract extract on. |
| | Pre op — OP — 1 Day — 1 Week — 1 Month — 3 Months |
| | FIGURE 1 - COHORT SCHEDULE |
| s. 1 s . | TI C. I C CUNTING C. II C C |
| Study Outcomes | The safety and performance of HMTIOL for the treatment of pre-ex st ng cornea |
| | ast gmat sm and aphak an subjects following cataract extraction with be |
| | character zed. |
| | Performance Outcomes: |
| | , |
| | <ol> <li>Post op MRCYL for eye mp anted w th HMTIOL</li> </ol> |
| | 2. Post op MRCYL pred ct on error for eye mp anted w th HMTIOL |
| | 3. Post op SEQ Pred ct on Error |
| | 4. UCDVA by study v s t |
| | 5. BCDVA by study v s t |
| | 6. IOL mer d an m sa gnment on the day of surgery |
| | 7. Rotat on of IOL mer d an from the day of surgery to 3 months, and |
| | between a adjacent v s ts |
| | a. Mer d an rotat on ≤ 5 |
| | b. Mer d an rotation < 10 |
| | c. Mer d an rotat on < 20 |
| | d. Mer d an rotat on < 30 |
| | e. Abso ute va ue of rotat on |
| | f. S gned va ue of the rotat on |
| | 8. Reduct on n cy nder power of eye mp anted w th HMTIOL ( n |
| | D opters) |
| | a. Abso ute preop magn tude of K (or tota cornea cy nder) m nus |
| | the abso ute post op magn tude of MRCYL at the cornea p ane |
| | 9. Percentage reduct on n cy ndr ca power of eye mp anted w th |
| | HMTIOL |
| | a. Abso ute preop magn tude of K (or tota cornea cy nder) m nus |
| | the abso ute post op magn tude of MRCYL at the cornea p ane |
| | expressed as a percentage of the abso ute preop magn tude of |
| | K (or tota cornea cy nder) |
| | Safaty Outcomes |
| | Safety Outcomes: |
| | Preservat on of BCDVA |

**Document:** TDOC-0055987

Status: Effective

CLARV STA MED CAL


PROTOCOL CP 00004 REV 01

Effective Date: 24-Apr-2019

2. Rate of dev ce-re ated Secondary Surg ca Intervent on's (SSI's) other than opt c exchange or rotat ona adjustment of the HMTIOL 3. Dev ce def c ency 4. AEs rates **Inclusion Exclusion Criteria** Inc us on cr ter a \*both eyes do not need to 1. Adu t at east 22 years of age at the t me of consent be eligible 2. Must be w ng and ab e to return for schedu ed treatment and fo owup exam nat ons for up to 6 months study durat on 3. P anned remova of v sua y s gn f cant cataract (cort ca, nuc ear, poster or subcapsu ar, or a comb nat on) by manua phacoemu s f cat on cataract extract on 4. Pre-ex st ng cornea ast gmat sm n the study eye. Magn tude of ast gmat sm w th n the range of ava ab e tor c power 1.50, 2.25 and 3.00D at the IOL p ane, after adjust ng for Surg ca y Induced Ast gmat sm. 5. Target d optr c ens power w th n the range of 16 – 26D 6. Must be w ng to d scont nue contact ens wear for the durat on of the study and demonstrate refract ve stab ty pr or to b ometry and surgery **NOTE:** Due to potent a var ab ty of VA and MR outcomes fo ow ng gas permeab e (GP) contact ens wear, a subjects who have worn GP contact enses must comp ete the consent ng process, d scont nue wear for 3 weeks and exh b t a stab e Man fest Refract on (as ev denced by

Document: TDOC-0055987

**Status:** Effective


Effective Date: 24-Apr-2019

CLARV STA MED CAL

two MR eva uat ons at east 1 week apart resu t ng n  $\leq$ 0.50D MRSE d fference n the two refract ons) and Keratometry read ngs (as ev denced by two K read ngs at east 1 week apart resu t ng n  $\leq$ 0.50D d fference between the two read ngs) pr or to f na IOL ca cu at ons. S m ar y, any subjects who current y wear soft contact enses must a so comp ete the consent ng process, d scont nue wear for a m n mum of 1 week and return for repeat e g b ty test ng exh b t stab e MR and K read ngs. In add t on, a qua fy ng subjects must d scont nue contact ens wear n the study eye for the durat on of study part c pat on.

- 7. BCVA projected to be 0.2 LogMAR or ower (as determ ned by the med ca judgment of the Invest gator or measured by potent a acu ty meter / ret na acu ty meter (PAM / RAM) f necessary)
- 8. V sua symptoms re ated to cataract
- 9. Stab ty of the cornea has been demonstrated by keratometry
- 10. D ated pup s ze at east 7.0mm
- 11. Must be able to understand and provide informed consent themse ves or through a representative with a witness present on the IRB or EC approved Informed Consent Form (ICF)

#### Exc us on cr ter a

- 1. H story of any ntraocu ar or cornea surgery n study eye (nc ud ng refract ve)
- 2. Any type of cataract (e.g. traumat c, congenta, po ar) other than those noted n nc us on cr ter a
- 3. Pregnancy or actat on
- 4. Part c pat on n any other drug or dev ce c n ca tr a w th n 30 days pr or to enro ng n th s study and/or dur ng study part c pat on
- 5. Prev ous cornea based surgery (LASIK, PRK, LRI, etc.)
- 6. H story of any c n ca y s gn f cant ret na patho ogy or ocu ar d agnos s (e.g. d abet c ret nopathy, schem c d seases, macu ar degenerat on, ret na detachment, amb yop a, opt c neuropathy, etc.) n study eye that cou d a ter or mtf na postoperat ve v sua prognos s
- 7. H story of any ocu ar cond t ons which could affect the stablity of the IOL (e.g. pseudoexfollation, zonu ar days s, evident zonu ar weakness or dehiscence, etc.) in study eye
- 8. Any anter or segment patho ogy ke y to ncrease the r sk of comp cat ons from phacoemu s f cat on cataract extract on (e.g. chron c uve t s, r t s, r docyc t s, an r d a, rubeos s r d s, c n ca y s gn f cant cornea, Fuch's, or anter or membrane dystroph es, etc.) n study eye

Rev 01, 06 June 2016 


Status: Effective


Effective Date: 24-Apr-2019

| | 9. Any v sua y s gn f cant ntraocu ar med a opac ty other than cataract n |
|---|---|
| | study eye (as determ ned by the nvest gator) |
| | 10. Uncontro ed g aucoma n study eye (per Invest gator judgement) |
| | 11. Subjects with large refractive errors (hyperopia/myopia) of ax a or |
| | patho og c or g n that, n the op n on of the nvest gator, cou d |
| | confound outcomes |
| | 12. Uncontro ed system c d sease (e.g. d abetes me tus, act ve cancer |
| | treatment, menta ness, etc.) |
| | 13. Subject who, in the cinical judgment of the invest gator, is not suitable |
| | for part c pat on in the study for another c in call reason, as documented |
| | by the invest gator |
| | 14. Severe dry eye that, n the op n on of the nvest gator, wou d mpar the ab ty to obtan re ab e study measurements |
| | 15. Tak ng system c med cat ons that, in the opin on of the investigator, |
| | may confound the outcome or ncrease the intraoperative and post- |
| | operat ve r sk to the subject (e.g. Tamsu os n Hydroch or de – F omax) |
| | or other med cat ons including anticho inergics, a pha adrenergic |
| | b ock ng agents w th s m ar s de effects (e.g. sma pup /f oppy r s |
| | syndrome) |
| | D scont nuat on Cr ter a Dur ng Surgery |
| | 1. V treous oss pr or to use of the nvest gat ona dev ce |
| | Pos t ve poster or pressure prevent ng safe mp antat on of the ens system |
| | 3. Anter or chamber hyphema prevent ng v sua zat on of mp antat on |
| | 4. Any zonu ar or capsu ar rupture or capsu ar bag nstab ty |
| | 5. Intraoperat ve m os s prevent ng v sua zat on of f xat on features |
| | 6. Need for concom tant procedures (e.g. g aucoma surgery, LRI, RK, |
| | LASIK, etc.) |
| | 7. Subject who, n the c n ca judgment of the nvest gator, s not su tab e |
| | for part c pat on in the study for another c in cal reason, as documented |
| | by the invest gator |
| Planned Analyses | A eyes with attempted study ensimple antation will be included in the safety |
| | ana yses. The performance outcomes w be summar zed based on eyes |
| | mp anted with HMTIOL. A data summaries with be performed based on |
| | observed data; no mputation for missing cinical outcomes will not be |
| | performed. |
| | For cont nuous var ab es, |
| | mean, standard dev at on, med an, m n mum, and max mum w be prov ded. |
| l | |


Status: Effective


For categor ca outcomes, the counts and percentages of eyes with each categor caleve of outcome with be summarized.

The cumu at ve and pers stent adverse events w be summar zed at 3 months

For BCDVA and UCDVA, the number and percentages of eyes w th v sua acu ty of 20/20 or better 20/25 or better, 20/32 or better, 20/40 or better, and worse than 20/40 at each v s t w be summar zed.

The MRSE pred ct on error w be calculated for each eye (Section 8) and summar zed using statistics for continuous variables. The MRCYL prediction error (per cy inder power and vector analysis) will be derived for eye with HMTIOL and summar zed using statistics for continuous variables.

The

Effective Date: 24-Apr-2019

reduct on n MRCYL (abso ute power) and the percent reduct on n cy nder power w be derived for each eyes mp anted with HMTIOL. Reductions w be summarized using statistics for continuous variables. Additional vector analyses on MRCYL may be provided.

IOL rotat on w be derived for each eye from Day 0 (surgery) to postoperative v s ts. The statistics for continuous variables w be provided. The number and percentage of eyes with rotation of  $\leq 5$ , < 10, < 20, and < 30 w be calculated.


Status: Effective

CLARV STA MED CAL


Effective Date: 24-Apr-2019

#### 1.0 Introduction

Cataract surgery s a m n may nvas ve procedure designed to restore v s on with short recovery time. Advances in instrumentation and techniques over the past few decades have facilitated the enhancement in safety which eld owing for reproducible outcomes. While the serious adverse event rate remains low, selecting the right intraocular ensions (IOL) implications and typically nicrosections and typically nicrosections. This is referred to as residual refractive error (RRE) and typically nicrosections in nicrosections approximately 0.6 diopters (D)<sup>2</sup> of uncorrected focusing power. Furthermore, it is reported that current biometry measurements for selecting the correct IOL and subsequent surgical methods are associated with:

- 1. Up to 16% of pat ents undergo ng add t ona surg ca correct on to ach eve 20/20 unass sted v s on<sup>2</sup>.
- 2. Up to 55% of pat ents fa ng outs de of the r targeted postoperat ve refract on by at east 0.5D<sup>3,4,5</sup>.
- 3. Between 14 and 24% of surger es result in greater than 1 D of residual refractive error, when using manufacturer suggested constants<sup>3</sup>.
- 4. Up to 6% of pat ents exper ence un ntended and s gn f cant post-operat ve rotat on of a tor c IOL<sup>4</sup>.

  Rotat ons between 5-40 degrees have been observed and for every 1 degree of rotat on, 3% of the correct ve power of the tor c surface s ost.

Pat ents are frequent y sat sf ed w th the resu ts of the r cataract surgery and enjoy re at ve y qu ck recovery w th restorat on of v s on. However, as expectat ons have evo ved over t me, pat ents are demand ng the same degree of spectac e ndependence that other refract ve surger es such as LASIK prov de. Current y ava ab e opt ons to he p ach eve spectac e ndependence when RRE s present nc ude: contact enses, cornea mod f cat on (surgery or other), IOL exchange/man pu at on, or su cus p acement of a "p ggyback" IOL. These a ternat ves have s gn f cant m tat ons and r sks.

Comp cat ons due to contact enses are rare; however, contact ens nto erance and contact ens-re ated nfect ons could be ser ous and sight threatening. For some patients, contact ensiwear is contrained cated and they must resort to the use of spectacies. Eight patients in particular have difficulty handing contact enses.

If the patient is will not accept the additional cost and risks of a secondary procedure, the physician has more options; however, each of them poses als gnificant risk to the patient as out ined below.

<u>Corneal modifications</u> have been performed on tens of m ons of people across the world with some form of refractive surgery (e.g. LASIK). For example, not the U.S. (where the most extensive data exists) 11.5M Americans have had corneal refractive surgery and over the next two decades many wineed cataract surgery. LASIK increases the kellood for residual refractive error post cataract surgery due to inaccurate IOL power calculations with both ometry. There is hes tation among many ophthalmologists to repeat LASIK for RRE after cataract surgery because the FDA has not specifically evaluated the safety and effect veness of repeated LASIK in this setting. All their sks associated with the original LASIK procedure apply to retreatment, along with the increased potential for epithe all ingrowth, corneal ectasial and less robust nomograms for IOL selection for post cataract patients.

Furthermore, even for eyes that have not undergone pr or cornea refract ve surgery, the FDA has not spec f cay eva uated the safety and effect veness of cornea refract ve procedures (e.g., ast gmat c keratotomy, LASIK, PRK, etc.) to address RRE fo owing ensire pacement surgery, so the use of approved assers for this purpose in the U.S. is considered off-labe, and the risks are not we characterized. For example, it is unclear how optical aberrations that might be present with an IOL in place are increased by aberrations induced by cornea refractive procedures, how kelly cornea refractive procedures are to induce induce induced by carnea refractive procedures are to induce induced by carnea refractive procedures are to induce in the procedure of the procedures are to induce in the procedure of the procedures are to induce in the procedure of the

Rev 01, 06 June 2016 


Status: Effective

CLARV STA MED CAL


Effective Date: 24-Apr-2019

Furthermore, cornea based interventions do not address the root cause of RRE after cataract extraction (imprecise IOL power selection) and expose the patient to a new and independent set of possible adverse events. Thus, it would be desirable to be able to correct or modify the optical result without the need to irreversibly and unpredictably a tericorneal it issue following cataract extraction.

<u>Sulcus placement of a "piggyback" IOL</u> s a procedure that has not been eva uated for safety and effect veness by the FDA so the use of approved IOLs for this purpose in the U.S. s off-labe. Among the complications reported with this procedure are secondary pigment dispersion, it is regular ties, chronic in the triangle of the procedure are secondary pigment dispersion, it is regular ties, chronic in the triangle of triangle of triang

<u>IOL Exchange/Manipulation</u> n genera, s techn cay cha eng ng for the surgeon and poses an atrogen c r sk to ntraocu ar structures nc ud ng the ens capsu e, r s, and endothe um of the cornea. The capsu ar bag f broses weeks after IOL mp antat on creat ng a strong adhes on between the capsu e and the IOL. Man pu at on of the capsu ar bag to remove an IOL s the major r sk n th s sett ng and can damage the capsu ar bag nc ud ng poster or capsu ar rupture and capsu ar bag d s ocat on. The capsu ar bag cannot be repa red once damaged. Th s r sk ncreases over t me as the capsu ar bag adheres to the IOL and hapt cs. Even when IOL exchange s not required, man pu at on of tradit on a IOL's to rotate or center the optic introduces the r sk of capsu ar or zonu ar damage which can cause further ensints bit y and ensimal position. Thus, it would be desirable to be able to correct RRE without the need to remove the entire IOL particularly after capsular contraction or fibros s.

The C arV sta Harmon TM Modu ar IOL System s a CE-approved device designed for safe and easy post-operative adjustment of residual refractive error (RRE). The modular IOL concept will serve as a valuable addition to the armamentarium of cataract surgeons. The goal of this technology is to improve refractive (spheric and toric) outcomes and avoid the significant risks of secondary procedures currently being performed as standard practice to address RRE in an indirect manner. It is anticipated that this modular ensible provided in the focus of this study.

- 1. Post-operative correction of residual spherical refractive error Based on existing performance of conventional cataract surgery, researchers have concluded that refractive outcomes in normal eyes should be within 0.5D for 45% and within 1D for 85% of cataract cases<sup>5</sup>. This theoretical performance goal stifial substantially short of the real-world outcomes seen with corneal refractive surgery and which cataract patients and surgeons increasingly demand. As a consequence, secondary procedures to optimize visual outcomes following cataract surgery can be as high as 16% in some practices, particularly for premium ensipatients<sup>2</sup>.
  - Modu ar IOL techno ogy s ntended to d rect y mprove refract ve outcomes w thout the nherent r sk of a fu ens exchange or resort ng to the use of a cornea refract ve aser. W th the HARMONI™ des gn the spher ca opt c component s ntended to a ow exchange for a d fferent power opt c or adjusted to a gn w th the v sua ax s w thout extens ve man pu at on of the de cate capsu ar bag, thereby avo d ng the potent a for ntraocu ar (e.g., capsu ar and endothe a) trauma that s seen w th trad t ona IOL exchanges.
- 2. Post-operat ve correct on of rotat onaly displaced or off-axis toric ensigher energy 1 degree a toric IOL axis is off from the true postoperative axis of ast gmatism, there will be a 3.3% ossiof toric correction. Study data supporting a recent approval of a toric IOL (P930014/S045) showed that 6.7% of eyes underwent a secondary surgical intervention (SSI) in the form of IOL repositioning to resolve RRE. The HARMONI™ modular technology can be used to improve outcomes in patients where the toric ensights been displaced to an unintended position during the post-operative period. The HARMONI™ optical ows for adjustment to align with the ast gmatic merid an orivisual axis without man pulation of the base component thereby avoiding the potential for capsular traumal that is seen when toric IOLs are man pulated in the post-operative period.

The C arV sta Harmon <sup>TM</sup> Monofoca (non-tor c) Modu ar IOL System has been ava ab e s nce 2015. A tor c vers on, the C arV sta Harmon <sup>TM</sup> Tor c Modu ar IOL System (HMTIOL), has been recent y CE-approved.

Rev 01, 06 June 2016 


Status: Effective


#### 2.0 OBJECTIVES

The object ve of this study is to demonstrate the safety and performance of the HARMONI™ Modu ar Toric IOL in patients with pre-existing ast gmatism.

Effective Date: 24-Apr-2019

The spec f c object ves are:

- To ref ne the A-constant (ens constant) of the HMTIOL.
- To evaluate the refractive outcomes including ast gmatism correction with HMTIOL in primary cataract surgery.
- To eva uate ax a and rotat ona stab ty of the HMTIOL.

#### 3.0 STUDY DESIGN

#### 3.1 Description of the Study

This is a prospective, multi-center study being conducted at up to 10 investigative sites. A is test with have linst tutional Review Board (IRB) or Ethics Committee (EC) review and approval prior to recruit ng potential subjects. Up to 200 eighbeing eighbeing subjects with visually significant cataracts with undergo cataract extraction during participation. Approximately 20 eyes, a maximum of 30 eyes, with being eighbeing eighbeing subjects with the subject with the subject with the subject with the subject with the HMTIOL. Eyes with corneal ast gmatism that is within the dioptric range of the toric IOL (1.50, 2.25 and 3.00D at the IOL plane after adjusting for Surgically Induced Ast gmatism) with the manufaction with the subjects with the process of the subjects with the process of the subjects with the subjects with the process of the subjects with the subject with th

#### Fo ow up:

• 1 Day, 1 Week, 1 Month, and 3 Months fo ow ng cataract extract on.



F gure 2 - Cohort Schedu e

A subjects enro ed n th s study w be evaluated for 3 months fo owng cataract extract on (see Append x A – Schedu e of Assessments).

#### 3.2 STUDY POPULATION

After comp et ng the nformed consent process, subjects w be screened for part c pat on n the study.

#### 3.2.1 INCLUS ON CR TER A

1. Adu t at east 22 years of age at the t me of consent

Rev 01, 06 June 2016 


Status: Effective

CLARV STA MED CAL


Effective Date: 24-Apr-2019

2. Must be w ng and ab e to return for schedu ed treatment and fo ow-up exam nat ons for up to 6 month study durat on, per eye.

- 3. P anned remova of v sua y s gn f cant b atera cataract (cort ca, nuc ear, poster or subcapsu ar, or a comb nat on) by manua phacoemu s f cat on cataract extract on
- 4. Pre-ex st ng cornea ast gmat sm n at east 1 eye. Magn tude of ast gmat sm 0.75 to 2.50D of cornea ast gmat sm (w th n the range of ava ab e tor c power 1.50, 2.25 and 3.00D at the IOL p ane after adjust ng for Surg ca y Induced Ast gmat sm)
- 5. Target d optr c ens power w th n the range of 16 26D
- 6. Must be w ng to d scont nue contact ens wear for the durat on of the study and demonstrate refract ve stab typr or to b ometry and surgery

**NOTE:** Due to potent a var ab ty of VA and MR outcomes fo owng gas permeable (GP) contact ensine wear, a subjects who have worn GP contact enses must complete the consenting process, discontinue wear for 3 weeks and exhibit a stable Manifest Refraction (as evidenced by two MR evaluations at least 1 week apart resulting in  $\leq 0.50D$  MRSE difference in the two refractions) and Keratometry readings (as evidenced by two Kireadings at least 1 week apart resulting in  $\leq 0.50D$  difference between the two readings) prior to final IOL calculations. Similarly, any subjects who currently wear soft contact lenses must also complete the consenting process, discontinue wear for a minimum of 1 week and return for repeatle gibit by testing exhibit stable MR and Kireadings. In addition, a liquality ng subjects must discontinue contact lense wear in the study eye for the duration of study participation.

- 7. BCVA projected to be 0.2 LogMAR or ower (as determ ned by the med ca judgment of the Invest gator or measured by potent a acu ty meter / ret na acu ty meter (PAM / RAM) f necessary)
- 8. V sua symptoms re ated to cataract
- 9. Stab ty of the cornea has been demonstrated by keratometry
- 10. D ated pup s ze at east 7.0mm
- 11. Must be able to understand and provide informed consent themselves or through a representative with a witness present on the IRB or EC approved Informed Consent Form (ICF)
- 3.2.2 EXCLUS ON CR TER A PR OR TO SURGERY
  - 1. H story of any ntraocu ar or cornea surgery n study eye (nc ud ng refract ve)
  - 2. Any type of cataract (e.g. traumat c, congen ta , po ar) other than those noted n nc us on cr ter a
  - 3. Pregnancy or actat on

Rev 01, 06 June 2016 

Document: TDOC-0055987

**Status:** Effective

CLARV STA MED CAL


Effective Date: 24-Apr-2019

4. Part c pat on n any other drug or dev ce c n ca tra w th n 30 days pr or to enro ng n th s study and/or

dur ng study part c pat on

5. Prev ous cornea based surgery (LASIK, PRK, LRI, etc.)

6. H story of any c n ca y s gn f cant ret na patho ogy or ocu ar d agnos s (e.g. d abet c ret nopathy, schem c

d seases, macu ar degenerat on, ret na detachment, amb yop a, opt c neuropathy, etc.) n study eye that

cou d a ter or mtf na postoperat ve v sua prognos s

7. H story of any ocu ar cond t ons which could affect the stablity of the IOL (e.g. pseudoexfoliation, zonu ar

d a ys s, ev dent zonu ar weakness or deh scence, etc.) n study eye

8. Any anter or segment patho ogy ke y to ncrease the r sk of comp cat ons from phacoemu s f cat on

 $cataract\ extract\ on\ (e.g.\ chron\ c\ uve\ t\ s,\ r\ t\ s,\ r\ docyc\ t\ s,\ an\ r\ d\ a,\ rubeos\ s\ r\ d\ s,\ c\ n\ ca\ y\ s\ gn\ f\ cant$ 

cornea, Fuch's, or anter or membrane dystroph es, etc.) n study eye

9. Any v sua y s gn f cant ntraocu ar med a opac ty other than cataract n study eye (as determ ned by the

nvest gator)

10. Uncontro ed g aucoma n study eye (per Invest gator judgement)

11. Subjects w th arge refract ve errors (hyperop a/myop a) of ax a or patho og c or g n that, n the op n on of

the nvest gator, cou d confound outcomes

12. Uncontro ed system c d sease (e.g. d abetes me tus, act ve cancer treatment, menta ness, etc)

13. Subject who,  $\,$ n the c  $\,$ n ca  $\,$ judgment of the  $\,$ nvest gator,  $\,$ s not su tab e for part c pat on  $\,$ n the study for

another c n ca reason, as documented by the nvest gator

14. Severe dry eye that,  $\,$ n the op n on of the  $\,$ nvest gator, wou d  $\,$ mpa r the ab  $\,$ ty to obta n re  $\,$ ab e study

measurements

15. Taking systemic medications that, in the opin on of the investigator, may confound the outcome or increase

the ntraoperat ve and post-operat ve r sk to the subject (e.g. Tamsu os n Hydroch or de – F omax) or other

med cat ons nc ud ng ant cho nerg cs, a pha adrenerg c b ock ng agents w th s m ar s de effects (e.g. sma

pup /f oppy r s syndrome)

3.2.3 D SCONT NUAT ON CR TER A DUR NG SURGERY

1. V treous oss pr or to use of the nvest gat ona dev ce

2. Post ve poster or pressure prevent ng safe mp antat on of the ens system

3. Anter or chamber hyphema prevent ng v sua zat on of mp antat on

4. Any zonu ar or capsu ar rupture or capsu ar bag nstab ty

5. Intraoperat ve m os s prevent ng v sua zat on of f xat on features

6. Need for concom tant procedures (e.g. g aucoma surgery, LRI, RK, LASIK, etc.)


Status: Effective


7. Subject who, n the c n ca judgment of the nvest gator, s not su table for participation in the study for another c n cal reason, as documented by the invest gator

Effective Date: 24-Apr-2019

#### 3.3 STUDY VISITS

The t m ng and frequency of each assessment to be performed at each v s t, w be carr ed out accord ng to "Append x A – Schedu e of Assessments."

Procedures to be fo owed n order to carry out each nd v dua assessment, are under separate cover (See study spec f c Manua of Procedures).

In a nstances for those subjects with both eyes enrolled, if the first study eye and secondary eye post-operative assessments cannot be seen on the same day and both remain "in-window," the subject must return for a separate visit in order to maintain "in-window" status for both eyes throughout study participation.

#### 3.3.1 PRE-OPERAT VE V S T - SCREEN NG/BASEL NE (DAY -90 TO DAY 0)

After providing informed consent (see Section 4.1), prospective subjects with be screened to determine whether they meet enrol menticriteria. Demographic information, relevant ocular history, and current ocular medication use with being considered enrolled. If a criteria are met, the subject with being considered enrolled, IOL calculation completed to determine appropriate HMTIOL power, and the subject scheduled for surgery.

#### 3.3.2 Day 0 V s t (Cataract Surgery and IOL Implantation)

Record any changes in concom tant med cations and med call history, prepare the subject for surgery in the study eye (see Surgical Procedure Guide), and re-review inclusion/exclusion criteria to ensure subject stigual fies to participate.

The Invest gator w carry out the surg ca procedure and HMTIOL mp antat on as spec f ed in the Surg ca Procedure Manua and the following details who be captured in both Source Documents and eCRFs:

- Date of surgery
- Operat ve eye
- Inc s on ocat on and s ze
- Ophtha m c V scoe ast c Dev ce (OVD) used
- A med cat on used pre-, ntra-, and post-operat ve y (ophtha m c and system c)
- Mode, ser a number, and d opter of HMTIOL mp ant components
- Tor c IOL power and ax s or entat on
- IOL nject on dev ce

Once the subject s conf rmed stab e post-surgery, prov de IRB / EC approved post-operat ve nstruct ons and d scharge.

Record any AEs, adverse device effects (ADEs), unexpected adverse device effects (UADEs), or device deficiencies (DD) (see Sections 6.1.1, 6.1.2, 6.1.3, or 6.1.4 respectively) observed pre-, intra-, or post-operatively.


Status: Effective


In the event the subject s not mp anted w th the HMTIOL, the surgeon w provide the best care opt on to the patient, including mp anting a commercially available IOL.

Effective Date: 24-Apr-2019

In the event the subject s not mp anted w th an HMTIOL dev ce due to an intra-operative complication, the subject will be discontinued (see Section 4.5).

#### 3.3.3 Post-Operat ve V s ts (Days 1-60)

A subjects mp anted w tha study ensw be seen for 1 Day, 1 Week, 1 and 3 Month assessments as out ned n Append x A.

IN ADDITION, the second eye, fegbe and enroed n the study, wbe mp anted during this time period. It is recommended (at the final discretion of the Investigator), to complete this procedure as close to the 1 Week Visit (after first eye cataract extraction) as possible. Since second eye assessments wbe completed on the same schedule as the first eye assessments (see Appendix A – Table 1), this wall ow the subject further convenience in attending as many post-operative billiation assessment visits as possible.

The Invest gator w carry out the second eye surg ca procedure as spec f ed n the Surg ca Procedure Manua and the fo ow ng deta s w be captured n both Source Documents and eCRFs:

- Date of surgery
- Operat ve eye
- Inc s on ocat on and s ze
- Ophtha m c V scoe ast c Dev ce (OVD) used
- A med cat on used pre-, ntra-, and post-operat ve y (ophtha m c and system c)
- Mode, ser a number, and d opter of HMTIOL mp ant components
- Tor c IOL power and ax s or entat on
- IOL nject on dev ce

Once the subject s conf rmed stab e post-surgery, prov de post-operat ve nstruct ons and d scharge.

NOTE: A concom tant med cat on, AE, and SAE co ect on must be cont nued throughout the course of the study. Any outcomes result ng in unacceptable RRE (as determined between Investigator and Subject), can be addressed with spectacies, a contact lens, or surgical correction. Any PO surgical adjustments to address RRE (corneal refractive surgery, lens exchange, lens rotation, etc.) will be carried out as determined to be in the best interest of the subject. The course of treatment will follow the Investigators SOC and be collected as a concomitant procedure. If surgical correction of the RRE is performed during the investigation period, the refractive error prior to secondary surgery is reported as the final result.

#### 3.3.4 3 MONTH V S T (DAY 80-100)

Assessments w be completed as indicated in Appendix A – Tables 1 and 2. In the event the second eye is out of window at this visit, the subject w in return in-window to complete second eye assessments.

#### 3.3.5 UNSCHEDULED V S TS

If at any time during the study, outside of the above scheduled visits, the subject requests or the Investigator determines the subject should be assessed, an unscheduled visit may occur. Adverse events and concomitant Rev 01, 06 June 2016


Status: Effective

CLARV STA MED CAL


Effective Date: 24-Apr-2019

med cat ons w be recorded and assessments deemed necessary by the Invest gator should be performed on either or both eyes.

If a subject s seen for mutpevsts durng a given vst window, the data from a vst that sintended to meet the protocol requirements for the scheduled vst should be captured in the vst eCRF. Where such a determination cannot be made, the first vst within the scheduled vst window will be used for completion of the protocol required vst. If assessments are missing from that vst, however captured at subsequent vsts within window, those assessments can be collected as part of the protocol vst. In such a circumstance, the vst date will remain consistent with the first vst established within the vst window, per the scenario above. Any additional and applicable data captured and associated with the Study Eye will be captured as an Unscheduled Vst.

#### 3.3.6 M SSED V S TS

If a subject m sses any schedu ed v s t and cannot be seen pr or to the start of the next v s t w ndow, the v s t w be cons dered "m ssed."

#### 4.0 STUDY METHODS

Pr or to recru tment of any subjects into the study, review and written approva of the protocol and informed consent must be obtained from the Institutional Review Board (IRB) or Ethics Committee (EC) by each participating cinical site.

#### 4.1 INFORMED CONSENT

Informed consent must be obtained and documented in writing prior to the initiation of any study procedures. The subject (or the subject siegally authorized representative) must be a lowed sufficient time to thoroughly read (or have explained), the informed consent form. The Investigator or his/her designed should answer any questions that the subject/representative might have. If the subject agrees to participate in the study, (i.e. provides informed consent) the subject/representative must significant significant form. The witness and the Investigator must also significant forms on the subject/representative. If applicable, it will be provided in a certificant forms at on of the local anguage. As part of the consenting process, the subjects will be informed of the right to treatment for any injuries related to the study. Any and a such treatment if necessary, will be paid for by the Sponsor to the extentitive since the subject's healthcare coverage (subject to local ethics committee approval). Completion of the consenting process as we can still date of the subject's signature on the informed consent form should be noted in the subject's medical chart.

Subjects who complete the informed consent process will be screened for eightly. Screened subjects will be recorded on site-specific screening logs and once they are determined as being eighbe, they will be enrolled into the study and an HMTIOL order placed with the Sponsor finecessary. All eighbe subjects will receive a stipend to attend scheduled study visits as an allowance for food, time, and trave expenses.

# 4.2 ASSIGNMENT OF SUBJECT IDENTIFICATION

A un que and sequent a subject dent f cat on number (ID) w be assigned at screening and never dup cated for another subject. This ID w be used on a study-related documents. To maintain confident a ty, the subject's name w not be recorded on any study document other than the informed consent form.

Rev 01, 06 June 2016 


Status: Effective


#### 4.3 SCREEN FAILURE

A record of screen fa ures and the reasons for the screen fa ures w be recorded in the subject source documents and captured in the eCRF for summary.

Effective Date: 24-Apr-2019

#### 4.4 SUBJECT COMPLETION

The subject has completed the entire study when the HMTIOL has been implanted and the Sponsor receives completed electronic Case Report Form (eCRF) documentation for a visits and a Study Exit eCRF. Subjects who require further follow-up for an AE will be followed according to Section 6.3.4.

A Study Ex t eCRF must be comp eted for a subjects who comp ete the c n ca nvest gat on.

#### 4.5 Subject Discontinuation

A subject MUST be d scont nued pr or to the f na study v s t for any of the fo ow ng reasons:

- Death
- Subject s enro ed and schedu ed for surgery but s not mp anted w th an HMTIOL n at east one eye
- Surg ca comp cat on(s) unre ated to the nvest gat ona dev ce prevent ng the mp antat on of the HMTIOL ( .e. capsu orhex s tear, zonu ar rupture, ev dent zonu ar weakness or deh scence, poster or capsu ar rupture, v treous oss, poster or capsu ar p aque, s gn f cant detached Descemet's membrane, s gn f cant anter or chamber b eed ng, r s ncarcerat on or damage, cornea endothe a touch, unsuccessfu / ncomp ete phacoemu s f cat on, hapt c and/or opt c damage/hapt c amputat on)
- Exp antat on of the HMTIOL System

If the study ens s exp anted, one postoperat ve v s t shou d be comp eted to record best-corrected d stance v sua acu ty (BCDVA) before the subject s d scont nued.

Subjects who withdraw from the study will be asked to complete procedures out ned in the 3 Month Visit (f withdrawn prior to that visit). Subjects who are terminated due to an AE will be followed, if possible, at least untiresolution or stabilization of the AE. Subject withdrawais will be documented clearly on the source document and applicable eCRF.

Pr or to d scont nu ng a subject, every effort shou d be made to contact the subject, schedu e a f na study v s t, and obta n as much fo ow-up data as poss b e. Adverse events w be fo owed as descr bed n Sect on 6.3.4. D scont nued subjects shou d be fo owed outs de of the study protoco accord ng to the Invest gator's norma postoperat ve standard of care.

A Study Ex t eCRF must be comp eted for a subjects who d scont nue from the c n ca nvest gat on.

#### 4.6 LOST TO FOLLOW UP

Subjects who m ss the r 3-month v s t, as defined by the v s t w ndows and cannot be contacted, may be considered ost to fo ow-up. A fo ow-up attempts w be documented and kept w th the subject's source documentation, and the app cable eCRFs w be completed.

Rev 01, 06 June 2016 


Status: Effective

CLARV STA MED CAL


Effective Date: 24-Apr-2019

Subjects that vo untar y w thdraw consent after mp antat on w th the HMTIOL w be considered Lost to Fo ow-Up and an Ex t Form w be completed.

#### 4.7 STUDY COMPLETION

C arV sta w not fy the Invest gators when to contact the IRB / EC to announce study comp et on at the s te.

#### 4.7.1 EARLY STUDY TERM NAT ON

C arV sta has the r ght to term nate th s study at any t me. Reasons for term nat ng the study may nc ude, but are not m ted to, the fo ow ng:

- The nc dence or sever ty of adverse events in this or any ongoing studies involving the same technology (flappicable), indicates a potential health hazard to subjects
- · Subject enroment sunsat sfactory
- Data record ng s naccurate or ncomp ete.

In the event of premature study term nat on, appropr ate not f cat on w be given to the Invest gators, IRB / ECs, and regulatory bodies as applicable. In addition, ClarV sta (or designee) w instruct a linvest gators to discontinue dispensing study materials or treatments, will ensure a subjects complete appropriate for ow-up, and will arrange study closeout visits at each site as appropriate.

#### 4.8 CONCOMITANT THERAPIES

#### 4.8.1 CONCOM TANT MED CAT ON

Concom tant med cat ons are any prescription drugs used by a subject until conclusion of study participation. Any medication the Investigator deems in the best interest of the subject, is acceptable to prescribe or administer. However, any and a lare to be recorded in both the Concomitant Medication source document and eCRF as we last the reason for use (indication). An AE is to be reported and/or recorded as appropriate (see Section 6.0).

#### 4.8.2 CONCOM TANT PROCEDURES

A concom tant procedure s any nvas ve or non-nvas ve ocu ar or per-ocu ar procedure that takes p ace dur ng study part c pat on and w be captured n both the Concom tant Procedure Source Document and eCRF. The fo ow ng are examp es of two such procedures:

- Any PO surg ca adjustments ( .e. cornea refract ve surgery, ens exchange, ens rotat on, etc.)
- Neodym um: Yttr um-a um num-garnet (Nd:YAG) procedure to treat Poster or Capsu e Opac f cat on (PCO), f necessary. Th s w be sted as "Nd:YAG Capsu otomy."

**Note:** Any Nd:YAG capsulotomy procedures prior to exit will be performed only in response to spontaneous subject complaints (i.e. not solicited by study personnel) of reduced Visual Acuity (VA) or glare that affects functional vision, which is associated with PCO or striae, and captured on the eCRF in SLE findings.

Rev 01, 06 June 2016 

**Document:** TDOC-0055987 **Version:** <sup>1</sup>

Status: Effective

CLARV STA MED CAL


Effective Date: 24-Apr-2019

An AE s to be reported and/or recorded as appropriate (see Section 6.0). Any procedure reported in the Concomitant Procedure eCRF must have a corresponding Indication sted in either the Ocular History or AE eCRF (Only exception: PCO – See Section 6.1 for further details).

#### 4.9 PROTOCOL DEVIATIONS

A protoco dev at ons, the date of dev at on, and reason w be documented in the Source Document and eCRF. A dev at ons w be categor zed as either major or minor in the following manner:

#### Major:

- Dev at ons mpact ng subject safety (e.g. e g b ty)
- Dev at ons impacting subject rights (e.g. consent)
- Dev at ons impacting data integrity (e.g. instrumentation, masking)

#### M nor:

• A other dev at ons (e.g. out of w ndow v s ts, m ssed data po nt, etc.)

A major dev at ons must be reported by the Invest gator to the Sponsor and IRB/EC mmed ate y. Subject assessments w cont nue per protoco for the durat on of p anned part c pat on un ess the dev at ons put the subject at r sk or the subject's cond t on requires that he/she be d scont nued from the study.

#### 5.0 STUDY MATERIALS

#### 5.1 DESCRIPTION OF TEST ARTICLE

| The HARMONI™ Modu ar Tor c Intrac | ocu ar Lens (HMTIOL) System | s des gned to a | ow safe exchange or | adjustment |
|---|---|---|---|---|
| of an IOL opt c after mp antat on. | | | | |
| | | • | | |

Document: TDOC-0055987


Effective Date: 24-Apr-2019

Status: Effective






#### 5.1.1 INSTRUCT ONS FOR USE

Refer to the Surg ca  $\,$  Gu de for a  $\,$  use and adm n strat on deta  $\,$  s.

#### 5.2 PACKAGING AND LABELING

A packag ng and abe ng w be consistent with the current study design. The abeing w nc ude at a min mum, the following:

- Sponsor name and address
- "For S ng e Use On y" statement (or equ va ent symbo)
- Ster ty symbo
- Storage temperature range requ rements or equ va ent (e.g. "Store at room temperature.")
- Exp rat on date
- Power des gnat on
- Un que ser a number
- Mode number

# 5.3 ACCOUNTABILITY

The Invest gator s respons be for keep ng accurate accountability records of the number of study enses received, dispensed, and returned to Sponsor. The study enses must be stored under the appropriate conditions in a secure area and are to be implicated only in subjects enrolled in the study, in accordance with the conditions specified in this protocol.


Status: Effective


Effective Date: 24-Apr-2019

A accountab ty records w nc ude the fo ow ng:

- Mode and ser a numbers
- Rece pt date
- · Quant t es rece ved
- In t a s (attr butab ty) of s te personne who received, d spensed, or returned study enses
- Date of use
- Subject and eye treated w th the study ens (by Subject ID and In t a s on y)
- Date returned to Sponsor
- Defect ve or damaged study dev ces

Per od ca y throughout the study and/or upon comp et on, the Sponsor (or designee) will rever ew and ver fy the Invest gator's accountability records. Following verification, and as directed by the Sponsor, a unused and explanted products must be returned to the Sponsor.

**Note:** In addition, any study lenses or components deemed defective, damaged, malfunctioning, or explanted <u>must</u> be retained by the site and returned to the Sponsor for evaluation. Under no circumstances are any components to be discarded or otherwise disposed of. If there is any question as to the applicability of this directive, consult the Protocol Contacts page of this protocol and discuss the situation with a Sponsor representative.

#### 5.4 OTHER MATERIALS

Add t ona mater as can be provided to sites for the duration of the study on an as-needed basis and may include:

- ETDRS ght box, g are source, and charts to perform the standard zed VA assessments descr bed in the Manua of Procedures
- Med ce njectors (for study ens nject on on y)
- S t amp camera

#### 6.0 Adverse Events

Safety assessments include adverse events/ser ous adverse events, and adverse device events. The reporting time period is from the time of consent through the last study visit (3 Month Visit post cataract extraction).

#### 6.1 Definitions

#### 6.1.1 Adverse Event (AE)

An AE s any untoward med ca event n a subject that does not necessar y have a causa re at onsh p to the study dev ce or protoco. AEs nc ude Adverse Dev ce Effects (ADEs). Cond t ons or d seases that are preex st ng and/or chron c but stab e shou d not be recorded on AE pages of the eCRF. S m ary, changes n a pre-ex st ng and/or chron c cond t on of d sease that are cons stent w th natura d sease progress on are NOT adverse events and a so shou d not be recorded on the AE pages of the eCRF.

Refer to Sect on 6.3.1 for instructions regarding events that require expedited reporting to the Sponsor and IRB/EC.


Status: Effective

CLARV STA MED CAL


Effective Date: 24-Apr-2019

Experience with cataract surgery and the implantation of IOLs has shown that some conditions can be considered normal or expected events following these procedures. The following may be considered normal or expected events after cataract surgery and only need to be reported as AEs as specified here:

- Ir ts (ce / f are) f treated onger than standard post-operative regimen or fit recurred after complete resolution
- Pers stent Cornea Stroma Edema (f present at 1 Month)
- Increased IOP on y f med ca /surg ca ntervent on s required (i.e. med cation, paracentes s man pulation)
- BCDVA decrease of 10 or more etters (2 nes) from any previous visit not secondary to any under ying condition present at time of enrol ment
- Any expected post-operative ocu ar event requiring a change in standard postoperative medication regimen

Note: PCO is not to be reported as an AE, as per ISO 11979-7:2014.

**Note:** The HMTIOL is designed for safety and ease of optic exchange and rotational adjustment post-primary cataract surgery. Optic exchange and optic rotation to refine refractive outcomes are not to be reported as AE's.

Part cu ar attent on shou d be pa d to ensure t me y and accurate report ng of any of the fo ow ng cataract surgery re ated events:

- Endophtha m t s
- Capsu ar njury
- V treous oss
- Macu ar edema
- Ret na detachment
- Lens d s ocat on
- Moderate to severe cornea edema
- Pup ary b ock / ang e c osure
- Hypopyon or hyphema

#### 6.1.2 Adverse Dev ce Effect (ADE)

An ADE s any untoward or un ntended effect, event, or response surround ng and w th a causa re at onsh p w th the use of a med ca dev ce. This definition may include any event resulting from insufficiencies or nadequacies in the instructions for use or the deployment of the device or other device maifunctions. This definition includes any event that is a result of a user error and any event that affects a user of the device (i.e. caregiver, bystander, etc.).

#### 6.1.3 UNANT C PATED ADVERSE DEV CE EFFECT (UADE)

A UADE s any ADE, which is unantic pated and poses air skito health or safety, or any if e-threatening problem or death caused by or associated with a device, if that effect, problem, or death was not previously identified in nature, severity or degree of incidence (see Investigator Brochure [IB]). UADEs also include any


Status: Effective


unant c pated s ght-threaten ng events and any other unant c pated ser ous prob em assoc ated w th a dev ce that re ates to the r ghts, safety, or we fare of subjects.

Effective Date: 24-Apr-2019

#### 6.1.4 DEV CE DEF C ENC ES (DD)

A Dev ce Def c ency (DD) s a fa ure of the dev ce to meet ts performance spec f cat ons or expectat ons, or otherw se not perform as intended. This can include either a maifunction or damage to the device or any part thereof, regard ess of the source of maifunction or damage, including user error, and regard ess of the presence of injury (or ack thereof) to subject, user, or bystander.

#### 6.2 AE EVALUATION

AEs exper enced in this study may be associated with the study device (i.e. ADE) or the study protocol as demonstrated in the following non-exhaustive is to flexamples:

#### Study Dev ce (ADE)

- IOL d s ocat on
- Exp ant due to hapt c break/damage
- Exp ant due to base and/or opt c damage

#### Study Protoco

- A erg c react on to d at ng drops
- Lens remnants fo ow ng surgery
- Capsu ar tear dur ng surgery to mp ant study dev ce

#### 6.2.1 EVALUAT ON

A AEs w be eva uated for and by the fo ow ng cr ter a:

- C ass f cat on (SAE, AE, ADE or comb nat on)
- D agnos s (or descr pt on f ADE)
- Sever ty
- Re at onsh p (Causa ty) to study protoco or dev ce
- Outcome
- · Treatment or act on taken

#### 6.2.1.1 CLASSIFICATION

When eva uat ng AEs, the Invest gator must determ ne f the event s ser ous us ng the fo ow ng gu de nes:

A Serious Adverse Event (SAE) s any AE (ocu ar or non-ocu ar) that:

- resu ts n death
- resu ts n ser ous njury, def ned as:
  - fe-threaten ng
  - permanent mpa rment of a body funct on (e.g. b ndness) or structure


Status: Effective


 necess tates med ca or surg ca ntervent on to prevent permanent mpa rment of a body funct on or permanent damage to a body structure, or

Effective Date: 24-Apr-2019

- resuts na potent a ysght-threaten ng cond ton
- s a ma funct on that m ght cause or contr bute to a ser ous njury or death f t were to recur
- requires in-patient hospitalization or prolongation of existing hospitalization, or
- eads to feta d stress, feta heath, a congenta abnorma ty, or b rth defect

\*Hosp ta zat on s a criter on for assessment of ser ousness. Hosp ta zat on in the absence of a medical AE s not in itself an AE. For example, the following reports of hosp ta zation without a medical AE should not be considered either serious or an AE:

- adm ss on for treatment of a pre-ex st ng cond t on not assoc ated w th the deve opment of a new AE or
  w th worsen ng of the pre-ex st ng cond t on (e.g. for work-up of pers stent pretreatment ab abnorma ty)
- soc a adm ss on (e.g. subject has no p ace to s eep)
- adm n strat ve adm ss on (e.g. for year y phys ca exam)
- opt ona adm ss on not assoc ated with a worsening of a pre-existing condition (e.g. elective cosmetic surgery or elective surgery for pre-existing repair of the Achiles tendon [which had not worsened while on study])
- hosp ta zat on for adm ss on w thout a med ca AE

NOTE: For the purposes of this protocol, any UADE will be considered an SAE.

#### 6.2.1.2 DIAGNOSIS OR DESCRIPTION

In a nstances, t s preferable to report a AEs and SAEs by diagnosis rather than a sign or symptom if possible. This may necess tate the revision of a previously reported AE or SAE as more information is obtained.

#### 6.2.1.3 SEVERITY

When evaluating AEs, the Investigator must determine the severity of symptoms using the following guide nes:

- M d: Subject awareness of a s gn or symptom that s eas y to erated, requires no treatment, and does not interfere with the subject's daily activities
- Moderate: Subject awareness of a s gn or symptom which may be a low level of concern to the subject and may interfere with daily activities, but can be relieved by s mple therapeutic care
- Severe: A s gn or symptom that interrupts the subject's daily activity and requires systemic therapy or other treatment

#### 6.2.1.4 RELATIONSHIP (CAUSALITY) TO STUDY DEVICE OR STUDY PROTOCOL

When eva uat ng AEs, the Invest gator must eva uate the re at onsh p of the event to the study dev ce and study protoco, us ng the fo ow ng gu de nes:

Rev 01, 06 June 2016 


Status: Effective


• Not Re ated: AEs which are clearly and incontrovert by due to causes other than the study device or study protoco (e.g. concomitant disease, etc)

Effective Date: 24-Apr-2019

- Re ated: AEs which are feit with a reasonable degree of certainty to be related to the study device or study protoco
- Unknown: Adverse events for which a connection with the study device or study protocol cannot be ruledout with certainty, or not enough information is available to assess the relationship

#### 6.2.1.5 OUTCOME

The c n ca outcome of an AE w be categor zed as fo ows:

- Reso ved w thout seque ae
- Reso ved w th seque ae (spec fy)
- Ongo ng ( .e. cont nu ng at t me of study d scont nuat on)
- Death

#### 6.2.1.6 TREATMENT OR ACTION TAKEN

Treatment or Act on Taken w be categor zed as fo ows:

- None
- Med ca Intervent on (spec fy on Concom tant Med cat on Source and eCRF)
- Surg ca Intervent on (spec fy on Concom tant Procedure Source and eCRF)
- Other (spec fy)

#### 6.3 REPORTING

#### 6.3.1 ON-S TE EXPED TED REPORT NG

The Invest gator s ob gated to report the fo ow ng to the Sponsor w th n 24 hours of becom ng aware of the event to ensure the safety of a part c pants n the study and to meet regulatory reporting requirements:

- A SAEs, regard ess of re at onsh p to study dev ce or study protoco ut z ng the SAE/ADE Report Form
- A AEs determ ned to be re ated to the study dev ce (ADEs or UADEs) ut z ng the SAE/ADE Report Form
- A HMTIOL exp ants (consult Medical Monitor is sted on Protoco Contacts page prior to explant, if possible)
- A Dev ce Def c enc es (DD) ut z ng the DD Report Form

Refer to the Protocol Contacts page for appropriate Sponsor contact to report the above events.

NOTE: Any explanted HMTIOL devices, exchanged HMTIOL optics, or any components of the HMTIOL System presenting a deficiency or malfunction are to be retained by the site until collected by the Sponsor. Under no circumstances are they to be destroyed or otherwise discarded.

When report ng these events to the Sponsor, the s te should forward any support ng documents a ong with the appropriate reporting form and complete the corresponding eCRF, if applicable. Sites must also report applicable events to the reviewing IRB/EC per its established reporting procedures.


Status: Effective


#### 6.3.2 OFF-S TE SAE REPORT NG

As a mut center c n ca tra, the Invest gators may receive "off-site" reports (e.g. an SAE Report). These are Sponsor reports of SAEs which occurred at other sites for the same tra, or in different trass using the same test article, that met the criteria for reporting. These should be reported to the reviewing IRB per their established reporting procedures.

Effective Date: 24-Apr-2019

#### 6.3.3 REPORT NG OF COMPLA NTS FOR ANC LLARY MARKETED PRODUCTS

Any comp a nts, ma funct ons or s m ar events reated to anc ary marketed products used n this study should be reported by the Investigators in accordance with the reference information provided on the associated commercial packaging.

#### 6.3.4 Adverse Events and Ser ous Adverse Events at Subject Ex t

Ongoing SAEs and ADEs will be followed until resolution or no further change in the condition is expected. Non-serious AEs that are ongoing at study exitivistic upon discontinuation from the study will be followed per the Investigator's standard of care. Documentation in the eCRF of this follow-up is not required a though subject care should continue as appropriate.

#### 6.4 SAFETY MONITORING AND REVIEW

A reported AEs w be reviewed on a weekly basis and assessed for trending and causality to study device or procedure ADEs, UADEs, DDs, and SAEs w be reviewed upon receipt of expedited reporting (Section 6.3.1). Any unexpected trends or events w necessitate careful review and assessment of any change in the risks associated with participation or study continuation.

f an event occurs affect ng a sub ect's r sk of part c pat on, Off S te Report ng (Sect on 6 3 2) w be ut zed to update s tes and the RB(s) / EC(s) f the safety prof e of the event prov des for the cont nuat on of the study, nformed Consent Forms w be rev sed as necessary to ensure sub ects' consent to cont nue part c pat on g ven the known rev sed r sks

As out ned in Section 4.7.1, the Sponsor reserves the right to discontinue enrollment at any time

#### 7.0 STUDY OUTCOMES

#### 7.1 SAFETY OUTCOMES

Safety w be evaluated by assess ng the following:

- · Preservat on of BCDVA
- Rate of dev ce-re ated SSI's other than opt c exchange and rotat ona adjustment of the HMTIOL
- AE rates
- Dev ce def c enc es

#### 7.2 Performance Outcomes

- Ca cu at on of Standard error of the mean n ens power A-constant for ref nement
- 1 and 3 months MRCYL for eyes mp anted w th HMTIOL
- 1 and 3 months MRCYL pred ct on error for eyes mp anted w th HMTIOL
- 1 and 3 months MRCYL pred ct on error for eyes mp anted w th HMTIOL per vector ana yses


Status: Effective


Effective Date: 24-Apr-2019

- 1 and 3 months SEQ pred ct on error
- UCDVA by study v s t
  - o Percent of eyes that ach eve
    - 20/20 or better
    - 20/25 or better
    - 20/32 or better
    - 20/40 or better
    - Worse than 20/40
- BCDVA by study v s t
  - Percent of eyes that ach eve
    - 20/20 or better
    - 20/25 or better
    - 20/32 or better
    - 20/40 or better
    - Worse than 20/40
- IOL mer d an m sa gnment on the day of surgery
- Rotat ona of IOL mer d an at 1 day, 1 week, 1 and 3 months
  - Percent of eyes w th rotat on  $\leq$  5
  - o Percent of eyes w th rotat on < 10
  - o Percent of eyes w th rotat on < 20
  - Percent of eyes w th rotat on < 30</li>
  - o Abso ute va ue of rotat on
  - 0
- Reduct on n cy nder power of the eye mp anted w th HMTIOL (abso ute preoperat ve magn tude of cornea cy nder (K) m nus the abso ute postoperat ve magn tude of MRCYL at the cornea p ane)
- Percentage reduct on n cy ndr ca power of the eye mp anted w th HMTIOL (abso ute preoperat ve magn tude of cornea cy nder (K) m nus the abso ute postoperat ve magn tude of MRCYL at the cornea p ane, expressed as a percentage of the abso ute preoperat ve magn tude of tota cornea cy nder (K)).



#### 8.0 STATISTICAL METHODS

This is a study to evaluate the safety and performance of HTMIOL in subjects undergoing cataract surgery. In general, the analyses will be provided based on available data. The mean, standard deviation, minimum, and maximum will be prepared for the continuous clinical parameters, and counts and percentages will be presented for the categorical outcomes.

# 8.1 SAMPLE SIZE CALCULATION


Status: Effective


The samp e s ze of th s study s based on ref nement of A-constant (ens power constant). To reduce b as due to surg caltechnique, unusual eyes and differences in equipment (A scan, keratometer, etc.) data will be obtained from a sufficient number of eyes such that the standard error of the mean in ens power constant is ession than  $\pm 0.10$ mm (approximate y  $\pm 0.2$ D). A min mum of 20 to 30 eyes from each surgeon should be adequate to achieve the tolerance. Each included subject should have a post-operative uncorrected visual activity better than 20/40 to avoid inaccuracies in refraction.

Effective Date: 24-Apr-2019

This is a feasibility study and no hypothesis testing will be performed.

#### 8.2 Analyses Populations

Subjects that are screened but d squa f ed based on the preoperat ve and ntra-operat ve e g b ty cr ter a w be exc uded from the safety and performance data ana yses. However, the r reasons for the screen fa ure w be summar zed. The ana yses popu at ons are defined be ow.

#### 8.2.1 SAFETY POPULAT ON

The **Safety Population** not udes eyes with attempted study ensimply antation, (successful or aborted after contact with the eye). The intraoperative and postoperative AEs and DDs will be summarized based on the safety population.

#### 8.2.2 IMPLANTED-EYE POPULAT ON

The **Implanted-Eye** Popu at on cons sts of eyes w th successfu HMTIOL mp antat on. Since it is important to evaluate HMTIOL's effection a study eyes, sit is ample examination, intraoperative pressure (IOP), and distinct fundus examination (DFE) will be based on the implanted-eye population.

Add t ona y, the UCDVA, BCDVA, pred ct on error, and mer d an rotat on w be eva uated based on the mp anted-eye popu at on.

#### 8.2.3 PER PROTOCOL POPULAT ON

The **Per Protocol** (PP) Popu at on contains eyes with successful HMTIOL implantations during surgeries and do not have a major protocol deviation (such as improperly enrolled in the study or lens power calculation errors) and will be considered the primary population for the analysis of performance outcomes. The performance outcomes (UCDVA, BCDVA, and prediction error) will also be evaluated based on the per protocol population.

The protoco dev at ons w be categor zed pr or to the ana ys s.



Rev 01, 06 June 2016 

**Document:** TDOC-0055987


Effective Date: 24-Apr-2019

Status: Effective




#### 8.3 STATISTICAL METHODS

The data analyses will be based on the analysis populations described above. No imputation for missing data will be performed. The demographic data will be summarized based on study subjects.

For cont nuous outcomes, mean, standard dev at on, med an, m n mum, and max mum w be provided. For categorica outcomes, the counts and percentages of eyes with each categorica eve of outcomes w be summarized.

#### 8.3.1 SAFETY OUTCOMES

# 8.3.1.1 ADVERSE EVENTS AND DEVICE DEFICIENCIES

Adverse events and device deficiencies will be summarized at each study visit based on the safety population. The number and percentage of eyes reported with the 3-month cumulative and persistent adverse events will be calculated.



#### 8.3.2 Performance Outcomes

The performance outcomes w be ana yzed based on the Imp anted-eye Popu at on and PP Popu at on. The BCDVA w a so be summar zed based on the Best-case popu at on as suggested by ISO.




Status: Effective


8.3.2.2 UCDVA

The proport on of eyes w th UCDVA of 20/20 or better, 20/25 or better, 20/32 or better, 20/40 or better, and worse than 20/40 at each v s t w be summar zed at the preoperat ve and every postoperat ve v s ts.

#### 8.3.2.3 PREDICTION ERROR (PE)

The MRSE pred ct on error w be calculated at 3 months for each implanted eye as follows:

MRSE PE = Postoperative MRSE adjusted to 6 meters - MRSE TRRE (target residual refractive error)

The MRCYL pred ct on error w be calculated at 3 months for eyes implanted with HMTIOL as follows:

MRCYL PE = Postoperative MRCYL adjusted to 6 meters – MRCYL TRRE (target residual refractive error)

The MRCYL PE w a so be calculated based on the vector analysis approach for eyes implanted with the HMTIOL.

#### 8.3.2.4 MISALIGNMENT OF IOL MERIDIAN

The f na rotat ona mer d an of the IOL w be compared to the p anned post on. The absolute value of rotat on w be described by mean, med an, and max mum values.

8.3.2.5 ROTATION OF IOL MERIDIAN

The rotat on of IOL mer d an w be calculated for each eye from Day 0 to every postoperative visit. The descriptive statistics for continuous variables w be used to summarize the rotation angle at each visit. The absolute value of rotation w be described by mean, med an, and maximum values.

The number and percentage of eyes

Effective Date: 24-Apr-2019

w th rotat on  $\leq 5$  , <10 , <20 , and <30~ w  $\;$  be ca cu ated at each v s t.

8.3.2.6 REDUCTION IN CYLINDER POWER

Document: TDOC-0055987

Status: Effective


Effective Date: 24-Apr-2019

CLARV STA MED CAL

The reduct on n cy nder power w be calculated for each eye mp anted with the HMTIOL as follows:

Cylinder Power Reduction = absolute value of preoperative magnitude of corneal cylinder (K) – absolute postoperative magnitude of MRCYL at the corneal plane.

The percent reduct on n cy ndr ca power w be calculated for eyes with non-zero preoperative corneal cy nder as follows:

Cylinder Power % Reduction = Cylinder Power Reduction/ absolute value of preoperative magnitude of corneal cylinder  $(K) \times 100$ .

The descriptive statistics for continuous variables will be used to summarize these outcomes at each visit.

The vector ana yses (Eyde man<sup>11</sup>) based on the cy nder power and ax s w be performed.

#### 9.0 DATA MANAGEMENT

#### 9.1 DATA QUALITY ASSURANCE

A requested information must be entered on the eCRF and confirmable through source documentation. If an item is not available or not applicable, this fact should be clearly indicated.

Data w be entered into a computer database developed specifically for this trail. During the course of the trail, queries w be generated for data points that are potentially erroneous and require appropriate carification or correction.

#### 9.1.1 DATA MON TOR NG

Per od c mon tor ng (e ther remote and/or on-s te) w take p ace to ensure data integrity. Study mon tor ng nvo ves the following e ements:

C arV sta personne, or designee, may meet with invest gators prior to the initiation of the study in order to review the adequacy of the subject population, facilities, and equipment with respect to the needs of the study, and to familiar zeithe investigator and support staff with the study protocol.

C arV sta personne, or des gnee, may meet with the invest gators at the time enrollment is initiated in order to ensure that subjects are being properly selected, that the methods described in the study protocollare thoroughly understood by the invest gator, and that study data are being correctly recorded.


Status: Effective


C arV sta personne, or des gnee, may v s t the c n ca s te at any t me dur ng the course of the study to rev ew and/or co ect comp eted case report forms. Add t ona y, te ephone consu tat on w occur as necessary dur ng the course of the study to ensure the proper progress and documentat on of the study f nd ngs.

Effective Date: 24-Apr-2019

The study data w be carefuly protected, and masking ut ized to the extent possible, in order to prevent bias.

#### 9.2 Record Retention

The nvest gator sha maintain a subject records for whichever of the following periods is shorter:

- A per od of two years after the date on wh ch FDA approves the market ng of the dev ce
- A per od of f ve years after the date on which the results of the study are submitted to the FDA in support of the marketing of the device.

OR

• A per od equa to the m n mum required by the regional authority.

The Invest gator / S te must contact C arV sta as prov ded n the Protoco Contacts page pr or to d scard ng or d spos ng of any study re ated supp es or documents. The Sponsor reta ns the r ght to have a study documents sh pped (at Sponsor's expense) for arch va purposes, as an a ternat ve to d sposa.

#### 10.0 REFERENCES

- Joshua D. Ste n, MD. Ser ous adverse events after cataract surgery. Current Opinions in Ophthalmology 23 2012 May: 219-225.
- 2. Sverker Norrby, PhD. Sources of error n ntraocu ar ens power ca cu at on. *Journal of Cataract and Refractive Surgery* 34 2008 Mar: 368-376
- 3. Retz aff JA, Sanders DR, Kraff MC. Deve opment of the SRK/T ntraocu ar ens mp ant power ca cu at on formu a. *J Cataract Refrat Surg* 1990 May: 16; 333-340
- 4. L m LH, Lee SY, Ang CL. Factors affect ng the pred ctab ty of SRK II I pat ents w th norma ax a ength undergo ng phacoemu s f cat on surgery. Singapore Med J 2009; 50 (2) 120-125
- 5. Ga e RP, Sa dana M, Johnston RL et a . Benchmark standards for refract ve outcomes after NHS cataract surgery. *Eye 23*, no. 1 2009 Jan: 149-152.
- 6. Ar st odemou P, Cartwr ght NE, Sparrow JM, Johnston RL. Intraocu ar ens formu a constant opt m zat on and part a coherence nterferometry b ometry: refract ve outcomes n 8108 eyes after cataract surgery. *J Cataract Refract Surg* 2011; 37:50 62.
- 7. Evans, BJW. Monov s on: a rev ew. Ophthal. Physiol. Opt. 2007; 27: 417-439
- 8. Er ckson, D.B. & Er ckson, P. Psycho og ca factors and gender d fferences n the acceptance of monov s on. *Perceptual and Motor Skills*, 2000; 91:1113-1119.
- 9. Back AP, Ho den BA, H ne NA. Correct on of presbyop a w th contact enses: comparat ve success rates w th three systems. *Optometry & Visual Science*. 1989 Aug; 66(8): 528-25
- 10. Du To t R, Ferre ra, JT, Ne ZJ. V sua and Nonv sua Var ab es Imp cated n Monov s on Wear. *Optometry & Visual Science*. 1998; 75 (2): 119-125

Alcon - Business Use Only Effective Date: 24-Apr-2019


Status: Effective


11. Eyde man M, et a . Standard zed Ana yses of Correct on of Ast gmat sm by Laser Systems That Reshape the Cornea. J of Refract ve Surg. 2006; 22: 81-95.


Status: Effective


Effective Date: 24-Apr-2019





Document: TDOC-0055987

Status: Effective

Effective Date: 24-Apr-2019

Document: TDOC-0055987


Effective Date: 24-Apr-2019

Status: Effective

APPENDIX A - TABLE 1: SCHEDULE OF ASSESSMENTS

| | Pre-Op Visit <sup>1</sup> | | Op Visit | | Form 4 | Form 5 | Form 6 |
|---|---|---|---|---|---|---|---|
| | | First Eye | Second Eye<br>(if enrolled) | Form 3 | | | |
| Procedure/Assessment | Day -90<br>to -0 | Day 0 | Day 0 (+3-30 Days<br>from the first eye<br>surgery) | 1 Day Visit<br>(Day 1-2 from<br>Day 0 of the<br>eye) | 1 Wk Visit<br>(Day 7-14 from<br>Day 0 of the<br>eye) | 1 Mo Visit<br>(Day 30-60<br>from Day 0 of<br>the eye) | 3 Mo Visit<br>(Day 80-100<br>from Day 0 of<br>the eye) |
| Informed Consent | X | | | | | | |
| Demographics | Х | | | | | | |
| Med/Ophthalmic History | X | X | X | | | | |
| Eligibility <sup>2</sup> | X | X | X | | X | X | X |
| UCDVA <sup>3</sup> | X | | | X | ^ | | |
| Auto and Manifest<br>Refraction | Х | | | | X | X | X |
| BCDVA | X | | | | | X | X |
| Keratometry <sup>4</sup> | X | | | | | X | |
| Axial Length | Χ | | | | 0.0000000000000000000000000000000000000 | | |
| Anterior Chamber Depth | X | | | | | | |
| IOL/Toric Power Calculation <sup>5</sup> | X | | | | | X | X |
| Slit Lamp Examination | X | | | Х | X | | X |
| IOP | X | | | X | X | X | ^ |
| Pupil Size | X | X | X | | | 5 CALL CO. 10 CO | |
| Surgery / IOL implantation | | X | X | | | X | Х |
| IOL Rotational Stability <sup>6</sup> | | X | X | X | X | X | X |
| (VE HOLDENSHIP) | | | | X | X | ^ | - |
| | | | | | | | X |
| Dilated Fundus Exam | X | | | | | | |

<sup>&</sup>lt;sup>1</sup> All testing to be conducted on both eyes

<sup>&</sup>lt;sup>2</sup> Will include pregnancy test if applicable

<sup>&</sup>lt;sup>3</sup> If UCDVA is < 20/40, perform Pinhole (PH) vision

<sup>&</sup>lt;sup>4</sup> Measurements via biometry will be utilized for both calculations and data capture

<sup>&</sup>lt;sup>5</sup> To be reviewed and approved by the Sponsor

<sup>&</sup>lt;sup>6</sup> Rotational stability as assessed by Reading Center

Document: TDOC-0055987

Status: Effective


Effective Date: 24-Apr-2019



**Document:** TDOC-0055987


Effective Date: 24-Apr-2019

Status: Effective